CLINICAL TRIAL: NCT06993532
Title: Cross-Cultural Adaptation, Validity, and Reliability of the Turkish Version of the Trapeziometacarpal Arthrosis Symptoms and Disability Questionnaire
Brief Title: Validity, and Reliability of the Turkish Version of the Trapeziometacarpal Arthrosis Symptoms and Disability Questionnaire
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Halil Ibrahim ERGEN, Assist. Prof., University of Gaziantep
Other Study IDs: 2023/346
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Trapeziometacarpal Arthrosis
Keywords: Trapeziometacarpal arthrosis, cross-cultural adaptation, Turkish version, reliability, validity
MeSH Terms: interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trapeziometacarpal arthrosis group: Patients aged 18 years or older, with a diagnosis of TMC arthrosis were included in the study.
  Interventions: Other: Validity and Reliability

INTERVENTIONS:
Other: Validity and Reliability — The TASD questionnaire, the Thumb Disability Examination (TDX) questionnaire, the Visual Analogue Scale (VAS) for pain, as well as hand grip and pinch strength measurements using the Jamar® Hydraulic Hand Dynamometer and Jamar Hydraulic Pinch Gauge Dynamometer were employed to assess thumb function and muscle strength. The questionnaires were administered twice, with a 7-day interval, during which no medical or rehabilitation intervention was made that could alter the clinical condition of the patients.

SUMMARY:
To our knowledge, a Turkish version of the TASD questionnaire, frequently used for assessing TMC arthrosis worldwide, does not currently exist. Therefore, proper translation and cross-cultural adaptation of the tool are necessary for non-English speaking patients. This study aimed to develop the Turkish version of the TASD questionnaire, and to demonstrate its reliability and validity for use in patients with TMC arthrosis.

DETAILED DESCRIPTION:
The original TASD was translated into Turkish independently by a physiotherapist with expertise in hand research and proficiency in English, a healthcare professional, and English teacher with no healthcare background. Demographic data were collected, followed by administration of the TASD questionnaire, the Thumb Disability Examination (TDX) questionnaire, the Visual Analogue Scale (VAS) for pain assessment, and hand grip and pinch strength measurements using the Jamar® Hydraulic Hand Dynamometer and Jamar Hydraulic Pinch Gauge to assess thumb function and muscle strength. The questionnaires were administered twice, with a 7-day interval, during which no medical or rehabilitation intervention was provided that could alter the clinical condition of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older,
* Diagnosis of Trapeziometacarpal arthrosis

Exclusion Criteria:

* Surgery on the thumb and/or hand/wrist,
* Acute trauma to the thumb,
* Cognitive problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of Trapeziometacarpal arthrosis with individuals
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Trapeziometacarpal Arthrosis Symptoms and Disability Questionnaire | 7 days
  The TASD was developed by Becker et al. to evaluate symptom intensity, disability severity, and treatment effectiveness in individuals with TMC arthrosis

SECONDARY OUTCOMES:
Thumb Disability Examination Questionnaire | 7 days
  The TDX consists of 20 items organized into three subcategories, evaluating limitations in ADLs, pain severity, and patient satisfaction with thumb function
Power Grip Strength and Pinch Strength | 7 days
  Power grip strength (PGS) and pinch strength (PS) were measured using the Jamar® Hydraulic Hand Dynamometer and Jamar® Hydraulic Pinch Gauge, respectively.
Visual Analogue Scale | 7 days
  Pain intensity was assessed by asking the patient to rate their current pain on a 10 cm scale (0, no pain, 10, intolerable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
a decision has not been made yet.

REFERENCES:
- [Background] Becker SJ, Teunis T, Ring D, Vranceanu AM. The Trapeziometacarpal Arthrosis Symptoms and Disability Questionnaire: Development and Preliminary Validation. Hand (N Y). 2016 Jun;11(2):197-205. doi: 10.1177/1558944715627239. Epub 2016 Feb 3. PMID 27390563
- [Background] Karademir F, Ayhan Kuru Ç, Yakut Y (2022) Cross-Cultural Adaptation, Reliability and Validity of the Turkish Version of the Thumb Disability Examination (TDX) Questionnaire . IFSSH, IFSHT, FESSH Combined Congress (pp.548). London, Canada.
- [Background] de Souza Almeida VA, Fernandes CH, Meireles LM, Faloppa F, Ejnisman B, Cohen M. Translation and cross-cultural adaptation of "Trapeziometacarpal Arthrosis Symptoms and Disability-TASD" into Brazilian Portuguese. Adv Rheumatol. 2021 Oct 9;61(1):61. doi: 10.1186/s42358-021-00218-z. PMID 34627390